CLINICAL TRIAL: NCT03762291
Title: Multiple Myeloma Trial of Orally Administered Salmonella Based Survivin Vaccine
Acronym: MAPSS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Premal Lulla, Assistant Professsor, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-42712 MAPSS
Record Dates: First submitted 2018-09-11; First posted 2018-12-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: hematologic malignancy; malignant proliferation of plasma cells; MM
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CVD908ssb-TXSVN (Experimental): 3 different dosing schedules will be studied (3+3 design). At the beginning, patients will start on the lowest dose (1 of 3 different levels) of TXSVN. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 3 dose levels are studied. If the side-effects are too severe, the dose will be lowered or the TXSVN administrations will be stopped. Each patient will receive 2 vaccinations at the same dose, 2 weeks apart, according to the following dosing schedules: The administration will be oral.
  Dose Level 1
  Day 0: 2 x 10^5 cfu
  Day 14: 2 x 10^5 cfu
  Dose Level 2
  Day 0: 2 x 10^6 cfu
  Day 14: 2 x 10^6 cfu
  Dose Level 3
  Day 0: 2 x 10^7 cfu
  Day 14: 2 x 10^7 cfu
  Interventions: Biological: CVD908ssb-TXSVN

INTERVENTIONS:
Biological: CVD908ssb-TXSVN — TXSVN may activate the immune system which is the participants body's ability to fight disease, and help develop a response against cancer cells that express Survivin. Survivin has been safely targeted using immune cells, drugs or direct inhibitors in over 50 patients with cancers in published reports.
  Survivin belongs to the group of proteins known as tumor-associated antigens (TAAs). These are cell proteins that are specific to the cancer cell. They either are not found or are found in low levels normal cells in the human body. More than 90% of myeloma cancer cells have been shown to possess large quantities of Survivin.
  Other Names: TXSVN

SUMMARY:
Multiple myeloma patients will receive a cancer vaccine, called TXSVN that has been derived from the bacteria Salmonella. TXSVN is a weakened form of a live vaccine strain of the Salmonella bacteria (also known as the CVD908ssb strain) that has been genetically modified in the laboratory to produce a protein known as Survivin that stimulates an immune response in the body to the Survivin tumor antigen. CVD908ssb has been administered to over 80 healthy donors as a Salmonella vaccine in reported clinical trials. This trial intends to explore administration of this vaccine at a lower dose than what was tested in healthy individuals.

Survivin belongs to the group of proteins known as tumor-associated antigens (TAAs). These are cell proteins that are specific to the cancer cell. They either are not found or are found in low levels normal cells in the human body. More than 90% of myeloma cancer cells have been shown to possess large quantities of Survivin.

TXSVN may activate the immune system which is your body's ability to fight disease, and help develop a response against cancer cells that express Survivin. Survivin has been safely targeted using immune cells, drugs or direct inhibitors in over 50 patients with cancers in published reports.

TXSVN, the modified strain of CVD908ssb has not been tested in humans to this date. TXSVN is an investigational product not approved by the U.S. Food and Drug Administration.

The purpose of this study is to find the largest safe dose of TXSVN, to learn what the side effects are, and to see whether this therapy might help participants with multiple myeloma.

DETAILED DESCRIPTION:
The vaccine will be administered orally (by mouth) as a solution mixed with sodium bicarbonate. Approximately 10 minutes prior to receiving the vaccine, participants will take sodium bicarbonate pills to assist with the absorption of the vaccine. Participants may be pre-treated with acetaminophen (Tylenol) and diphenhydramine (Benadryl). Acetaminophen (Tylenol) and diphenhydramine (Benadryl) are given to prevent a possible allergic reaction to the vaccine. Participants will remain in the clinic for three hours after receiving the vaccine for monitoring.Two doses of TXSVN will be given two weeks apart. Participants disease will be assessed pre-treatment and then 6 weeks after the second treatment. All of the treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital.

In between the first and second treatments, and for 6 weeks after the last treatment, the investigators ask that participants not receive any other anti-cancer treatments such as radiation therapy or chemotherapy. If participants do receive any other therapies in-between the first and second treatment, then they will be taken off treatment and will not be able to receive the second treatment of cells.

This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose (1 of 3 different levels) of TXSVN. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 3 dose levels are studied. If the side-effects are too severe, the dose will be lowered or the TXSVN administrations will be stopped.

Before being treated, participants will receive a series of standard medical tests:

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurement of participants multiple myeloma by blood tests and bone marrow biopsy (when available).
* Measurements of participants tumor by routine imaging studies. The investigators will use the imaging study that was used before to follow the participants tumor: Computerized Tomography (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET/CT), skeletal bone survey. These studies will be done on a case-by-case basis at the discretion of the participants treating physician.
* Pregnancy test (using a blood sample) if the participants is a female who can have children.

Participants will receive standard medical tests when they are getting the vaccine and after:

* Blood tests to measure blood cells, kidney and liver function.
* Blood and stool cultures at 4 days after getting the vaccine and at least weekly for up to 8 weeks after treatment, to monitor shedding of the administered live vaccine.
* Measurement of the participants multiple myeloma by blood tests and/or bone marrow biopsy (when available). Imaging study (as decided by the participants treating physician) 8 weeks after the 1st vaccination.
* Participants will then come to the clinic every 3 months for the first year

To learn more about the way the vaccine is working in the participants body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before each vaccination, and weekly for eight (8) weeks after the participants first vaccination.

Study Duration: The participants active participation in this study will last for approximately one (1) year. The investigators will then contact the participants once a year for up to 4 additional years (total of 5 years follow-up) in order to evaluate the participants disease response long-term. While participants are being followed on study, investigators will collect information about the response to the vaccine (how well or not the participants multiple myeloma responds to the treatment) and any toxicities the participants may experience. This study will continue until it has completed enrolling subjects and all subjects have completed follow-up or have come off study.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient, greater than or equal to 18 yrs old regardless of sex, with a diagnosis of Myeloma after receiving at least two lines of conventional therapy which can include an autologous HSCT. If a patient has received an autologous or syngeneic SCT they must be greater than 90 days post-transplant
2. Patients with life expectancy greater than or equal to 6 weeks.
3. Pulse oximetry of greater than 90% on room air in patients who previously received radiation therapy to the chest. This is not required in patients who have not received radiation therapy to the chest in the past.
4. Patients with a Karnofsky score of greater than or equal to 50
5. Patients with bilirubin less than or equal to 2x upper limit of normal and Hgb greater than or equal to 7.0 (transfusion allowed).
6. AST less than or equal to 3x upper limit of normal.
7. ANC greater than 1000 at the time of vaccination and an ALC greater than 500.
8. Patients with a creatinine less than or equal to 2x upper limit of normal for age.
9. Patients should have been off other investigational therapy for one month prior to entry in this study.
10. Patients should be off anti-bacterial therapy for 14 days prior to vaccination
11. Patients should have been off conventional therapy for at least 1 week prior to entry in this study except immunomodulator drugs
12. Informed consent explained to, understood by and signed by patient. Patient given copy of informed consent.
13. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom. Females of child-bearing potential must be willing to utilize one of the more effective birth control methods during the study unless female has had a hysterectomy or tubal ligation.
14. Ability to swallow medications

Exclusion Criteria

1. Severe intercurrent infection.
2. Patients receiving greater than 0.5 mg/kg/day (prednisone equivalent) of systemic corticosteroids
3. Pregnant or breast feeding.
4. Grade II or higher nausea, vomiting or diarrhea.
5. History of allergy to prior vaccination with a Salmonella vaccine
6. HIV infection
7. Unable to tolerate Salmonella directed antibiotics
8. Household contacts who are immunocompromised, pregnant or under 2 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity (DLT) by CTCAE, v5.0 | 8 weeks
  Incidence of dose limiting toxicities (DLT) of CVD908ssb-TXSVN vaccine in patients with multiple myeloma.

SECONDARY OUTCOMES:
Overall response rate according to the modified International Myeloma Working Group (IMWG) Uniform Response criteria. | 8 weeks
  Overall response rate is defined as the proportion of subjects with best overall response of complete response (CR), stringent complete response (sCR), very good partial response (VGPR) or partial response (PR) according to the modified International Myeloma Working Group (IMWG) Uniform Response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Lulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No